CLINICAL TRIAL: NCT05119426
Title: An Open-label Effectiveness Study of a Typhoid Conjugate Vaccine in Kisantu, Democratic Republic of Congo (TyVECO) - Step 2: Typhoid Conjugate Vaccine (TCV) Mass-vaccination Campaign
Brief Title: Effectiveness of a Typhoid Conjugate Vaccine in DRC
Acronym: TyVECO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Vaccine Institute (Other)
Collaborators: Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other); University of Cambridge (Other); Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021-009
Record Dates: First submitted 2021-10-18; First posted 2021-11-15 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Typhoid Fever
Keywords: Typhoid conjugate vaccine; Vaccine effectiveness; Mass vaccination campaign; Democratic Republic of Congo (DRC)
MeSH Terms: conditions — Typhoid Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vi-TT (Experimental): Single dose of Vi-TT to children 9 months to <16 years of age
  Interventions: Biological: Vi-TT

INTERVENTIONS:
Biological: Vi-TT — Single dose of vaccine administered through a mass vaccine campaign to children between 9 months and <16 years of age. The campaign will emulate vaccine delivery as would be administered in a local mass vaccination campaign.
  Other Names: Typbar TCV

SUMMARY:
This is a prospective cohort evaluation of vaccine effectiveness of a single dose of Typbar-TCV® against symptomatic blood culture-confirmed typhoid fever when administered through a mass vaccination campaign to children 9 months to <16 years of age in Kisantu, DRC.

DETAILED DESCRIPTION:
This study is conducted in Kisantu, DRC and is comprised of a mass vaccination campaign of children aged 9 months to <16 years with a single dose of Typbar-TCV® and a concomitant surveillance study to assess the incidence of culture-confirmed typhoid fever in the population during a period of three years following vaccination. Safety events will be monitored for 30 minutes following vaccination for all participants. In a subset of age-eligible participants living in the study area, the investigators will assess local and systemic solicited adverse events/adverse reactions and unsolicited adverse events occurring within the first 7 days post-vaccination and unsolicited and serious adverse events within 28 days post-vaccination. A population census will be conducted at baseline to enumerate and characterize the population under study and demographic information will be collected to allow for minimization of potential sources of bias during analysis. An interim censuses and a census at study closure will be carried out to update population information.

The investigators hypothesize that the Typbar-TCV® vaccine is effective in large scale vaccination campaigns, thereby lowering the incidence of blood-culture confirmed typhoid fever in children. Lessons and experiences on vaccination feasibility and uptake will be important for informing TCV introduction across the African continent.

ELIGIBILITY:
Inclusion Criteria:

* Parent/guardian willing and able to provide informed consent; assent will be sought for participants between 12 and <16 years of age
* Resident of the defined study area, Kisantu Health Zone at the time of vaccination
* Age between 9 months and <16 years (i.e., ≤15 years and 364 days) on the day of vaccination

Exclusion Criteria:

* The participant has a known allergy to any of the vaccine components,
* Any medical reason perceived to increase risk to health posed by vaccination as judged by a medical professional
* Self-reported pregnancy in females greater or equal to 11 years of age who have reported menarche

Ages: 9 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48000 (Estimated)
Dates: Start 2022-02-11 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Direct vaccine effectiveness of Typbar-TCV® | 3 years
  Comparison of incidence of blood culture confirmed Salmonella Typhi infection in participants 9 months to <16 years of age vaccinated with a single dose of Typbar-TCV® delivered through a mass vaccination campaign and unvaccinated participants 9 months to <16 years of ageSalmonella Typhi isolated from blood specimens using conventional microbiological techniques

SECONDARY OUTCOMES:
Overall vaccine effectiveness of Typbar-TCV® | 3 years
  Comparison of incidence of blood culture confirmed Salmonella Typhi infection in all individuals 9 months to <16 years of age residing in clusters with lowest vaccine coverage (delineated virtually using GIS data) and all individuals 9 months to <16 years of age residing in clusters with highest vaccine coverage
Total vaccine effectiveness of Typbar-TCV® | 3 years
  Comparison of the incidence of blood culture confirmed Salmonella Typhi infection in vaccinated individuals 9 months to <16 years of age residing in clusters with highest vaccine coverage (delineated virtually using GIS data) versus unvaccinated individuals 9 months to <16 years of age residing in clusters with lowest vaccine coverage
Indirect vaccine effectiveness of Typbar-TCV® | 3 years
  Comparison of the incidence of blood culture confirmed Salmonella Typhi infection in unvaccinated individuals 9 months to <16 years residing in clusters with lowest levels of vaccine coverage (delineated virtually using GIS data) versus unvaccinated individuals 9 months to <16 years of age residing in clusters with highest levels of vaccine coverage
Safety profile of Typbar-TCV® | 28 days
  Proportion of participants developing local and systemic solicited adverse events/adverse reactions and unsolicited adverse events within the first 7 days post-vaccination in a subset of vaccinees and unsolicited and serious adverse events within 28 days post-vaccination
Feasibility of a single-dose Typbar-TCV® mass campaign in Kisantu, DRC | 3 years
  Descriptive report assessing both the scientific feasibility, including the ability of the study team to measure the above-named objectives, and operational feasibility, focusing on logistical aspects of the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Florian Marks, PhD, Principal Investigator — University of Cambridge; Octavie Lunguya, PhD, Principal Investigator — Institut National de Research Biomédicale
Locations (25):
- Democratic Republic of the Congo (25):
  - Cerphytoco, Kisantu, Bas-Congo Province
  - CS Cederi Madimba, Kisantu, Bas-Congo Province
  - CS Kavuaya, Kisantu, Bas-Congo Province
  - CS Kilenda, Kisantu, Bas-Congo Province
  - CS Kimuisi, Kisantu, Bas-Congo Province
  - CS Kinkonko, Kisantu, Bas-Congo Province
  - CS Kintanu Etat, Kisantu, Bas-Congo Province
  - CS Kipako, Kisantu, Bas-Congo Province
  - CS Kipasa, Kisantu, Bas-Congo Province
  - CS Kivuangi, Kisantu, Bas-Congo Province
  - CS Lemfu, Kisantu, Bas-Congo Province
  - CS Ngeba, Kisantu, Bas-Congo Province
  - CS Saint Pierre Boko, Kisantu, Bas-Congo Province
  - CS Yimbi, Kisantu, Bas-Congo Province
  - Gare, Kisantu, Bas-Congo Province
  - Kimayala, Kisantu, Bas-Congo Province
  - Nkandu 1, Kisantu, Bas-Congo Province
  - Nkandu 2, Kisantu, Bas-Congo Province
  - Nkandu 3, Kisantu, Bas-Congo Province
  - PS Kilemfu Nkanga, Kisantu, Bas-Congo Province
  - PS Kongo Nord, Kisantu, Bas-Congo Province
  - PS Ngombi Kinsambu, Kisantu, Bas-Congo Province
  - Site avancé de Kinsambamba, Kisantu, Bas-Congo Province
  - Unadic, Kisantu, Bas-Congo Province
  - Wete, Kisantu, Bas-Congo Province

IPD SHARING:
Plan to Share IPD: No
Sharing can be considered on a case-by-case basis considering the intended use and impact.